CLINICAL TRIAL: NCT05398328
Title: Effect of Personality Traits on Reporting Outcomes of Orthodontic Treatment
Acronym: OrthoPers
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rijeka (Other)
Responsible Party: Principal Investigator, Stjepan Spalj, Professor, University of Rijeka
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 2107-57-006-20-1
Record Dates: First submitted 2022-05-23; First posted 2022-05-31 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Malocclusion
Keywords: malocclusion; personality trait; quality of life
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: statistician will not be aware of group affiliation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- metal appliance + fixed retainer (Active Comparator): fixed metal appliance MBT 0.022'' slot in active phase followed by bonded wire retainer
  Interventions: Device: active metal appliance; Combination Product: retention fixed appliance
- esthetic appliance + fixed retainer (Experimental): fixed ceramic appliance MBT 0.022'' slot in active phase followed by bonded wire retainer
  Interventions: Device: active esthetic appliance; Combination Product: retention fixed appliance
- metal appliance + removable retainer (Active Comparator): fixed metal appliance MBT 0.022'' slot followed by removable clear termoplastic retainer
  Interventions: Device: active metal appliance; Combination Product: retention removable appliance
- esthetic appliance + removable retainer (Experimental): fixed ceramic appliance MBT 0.022'' slot followed by removable clear termoplastic retainer
  Interventions: Device: active esthetic appliance; Combination Product: retention removable appliance

INTERVENTIONS:
Device: active metal appliance — fixed metal labial orthodontic appliance MBT 0.022'' slot
  Arms: metal appliance + fixed retainer; metal appliance + removable retainer
Device: active esthetic appliance — fixed ceramic labial orthodontic appliance MBT 0.022'' slot
  Arms: esthetic appliance + fixed retainer; esthetic appliance + removable retainer
Combination Product: retention fixed appliance — fixed lingual metal retention appliance
  Arms: esthetic appliance + fixed retainer; metal appliance + fixed retainer
Combination Product: retention removable appliance — removable clear termoplastic retention appliance
  Arms: esthetic appliance + removable retainer; metal appliance + removable retainer

SUMMARY:
The study will monitor changes induced by orthodontic treatment and in the retention period, two years after the end of orthodontic treatment. The alignment of teeth, hygiene and gingiva will be assessed. Efficiency of two types of fixed appliances in active phase will be compared - esthetic and metal. Efficiency of two types of retention appliances in retention phase will be compared - fixed and removable.

The benefits of orthodontic treatment to be studied are aesthetic concerns, dental self-confidence, self-esteem, social contacts, psychological influences, and chewing limitation. The stability of personality traits, body image and perfectionism will also be analyzed, as well as the extent to which these dimensions modify the reporting of psychosocial effects of malocclusion treatment.

DETAILED DESCRIPTION:
The aim is to analyze:

1. the extent to which the type of device (metal / aesthetic) affects changes in quality of life (QoL)
2. whether the change in QoL is influenced by personality traits during therapy
3. long-term change in QoL and personality traits (before therapy, during, at the end and in retention for 2 years)
4. whether long-term QoL change is influenced by personality traits
5. dependence of relapse (incidence and intensity) on the type of retention appliance
6. change in QoL and personality trait depending on relapse
7. whether the change in QoL due to relapse is influenced by personality traits

ELIGIBILITY:
Inclusion Criteria:

- malocclusion with moderate or great need for orthodontic treatment (Index of Orthodontic Treatment Need grades >=3)

Exclusion Criteria:

- neurodevelopmental disorders, intellectual disability, oligodontia, congenital craniofacial anomalies, orofacial clefts

Ages: 13 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 120 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
irregularity of teeth | 48 months (start, 3 months, 1 year, 2 years, 1 year retention, 2 years retention)
  Little Irregularity Index - sum of displacement of contact points of frontal teeth (range 0-10 mm), higher score mean worse outcome
patient reported impacts of malocclusion | 48 months (start, 3 months, 1 year, 2 years, 1 year retention, 2 years retention)
  Malocclusion Impact Questionnaire with 17 aspects, each on 3-point scale (summary score on scale 0-51), higher score mean worse outcome
big five personality traits | 48 months (start, end of treatment, 1 year retention, 2 years retention)
  Big Five Inventory with 44 statements, each on 5-point scale, grouped into 5 traits: (extroversion (range 8-40), agreeableness (range 9-45), openness (range 10-50), conscientiousness (range 9-45) and neuroticism (range 8-40). higher score mean worse outcome

SECONDARY OUTCOMES:
normative orthodontic treatment need | 48 months (start, end of treatment, 1 year retention, 2 years retention)
  clinically assessed by using Index of Orthodontic Treatment Need - Dental Health Component with 5 grades, range 1=no/minor need - 5=very great need
esthetic treatment need | 48 months (start, end of treatment, 1 year retention, 2 years retention)
  assessed by using Index of Orthodontic Treatment Need - Aesthetic Component with 10 grades, range 1=no need - 10=very great need
retainer failure | 24 months
  number of railures of retainer in retention phase, nigher number indicates worse outcome
limitations of jaw function | 48 months (start, 3 months, 1 year, 2 years, 1 year retention, 2 years retention)
  Jaw Function Limitation Scale with 6 items on 11-point scale (0=no limitation-10=extreme limitation), average score, higher score indicates worse outcome
self-esteem | 48 months (start, 3 months, 1 year, 2 years, 1 year retention, 2 years retention)
  Rosenberg Self-Esteem Scale with 10 items on 5-point scale (1=not at all-5=very much), summary score on scale 5-50, higher score indicates better outcome
body image | 48 months (start, end of treatment, 1 year retention, 2 years retention)
  4 items on 5-point scale (1=not at all-5=very much), total score 4-20, higher score indicates better outcome
perfectionism | 48 months (start, end of treatment, 1 year retention, 2 years retention)
  35 items on 5-point scale (1=completely disagree-5=completely agree), range 29 - 145, higher score indicates better outcome
psychosocial imapcts of dental esthetics | 48 months (start, 3 months, 1 year, 2 years, 1 year retention, 2 years retention)
  23 items on 5-point scale (0=not at all-4=very much), grouped in 4 dimensions - aesthetic concern (range 0-12), dental self-confidence (range 0-24), social influence (range 0-32), psychological influence (range 0-24)), higher score means worse outcome for psychological influence, social influence and aesthetic concern, while in dental self-confidence higher score indicates better outcome
wite spot lesions of enamel | 48 months (start, 3 months, 2 years, 1 year retention, 2 years retention)
  number of teeth with enamel defects, scale 0-32, higher number means worse outcome
oral hygiene | 48 months (start, 3 months, 2 years, 1 year retention, 2 years retention)
  Silness-Loe index and Williams modification for subjects in orthodontic treatment on a scale from 0=no biofilm to 3=a continuous line greater than 1mm, mean of all measurement site is used, range 0-3, higher score means worse outcome
extent of gingivitis | 48 months (start, 3 months, 2 years, 1 year retention, 2 years retention)
  Full Mouth Bleeding Score on a scale 0-100%, higher percentage means worse outcome
gingival enlargement | 48 months (start, 3 months, 2 years, 1 year retention, 2 years retention)
  Seymour index (thickness (scale 0=normal-2=thickening >=3mm) + proportion of tooth crown coverage (scale 0=normal-3=papilla involving .2/3 of adjacent tooth crown half) on frontal teeth vestibular and oral in both jaws; scale 0-100), higher score means worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Stjepan Spalj, PhD, Principal Investigator — Sveuciliste u Rijeci
Locations (1):
- University of Rijeka, Faculty of Dental Medicine, Rijeka, Croatia

IPD SHARING:
Plan to Share IPD: Yes
Data obtained through this research may be provided to qualified researchers with academic interest in orthodontic treatment. Data or samples shared will be coded, with no PHI included. Approval of the request and execution of all applicable agreements (i.e. a material transfer agreement) are prerequisites to the sharing of data with the requesting party.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data requests can be submitted starting 9 months after article publication and the data will be made accessible for up to 24 months. Extensions will be considered on a case-by-case basis
Access Criteria: Access to trial IPD can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a Data Sharing Agreement (DSA). For more information or to submit a request, please contact princial investigator Stjepan Spalj.